CLINICAL TRIAL: NCT00586378
Title: Ovatio DR and VR Implantable Cardioverter Defibrillators Post-approval Study
Acronym: Post-Ovatio
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ELA Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITAC05
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-03

CONDITIONS: Sudden Cardiac Death
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Ovatio DR and Ovatio VR — implantable cardioverter defibrillator
  Other Names: Ovatio DR 6550 Dual-Chamber ICD; Ovatio VR 6250 Single-Chamber ICD

SUMMARY:
The purpose of this post-approval study is to confirm the safety and effectiveness of Ovatio DR and VR ICDs

ELIGIBILITY:
Inclusion Criteria:

* Candidates will come from the investigator's general ICD population who meet any of the accepted indications for an ICD implant according to the "ACC/AHA/ESC 2006 Guidelines for Management of Patients With Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death" (Zipes et al., JACC Vol. 48, No. 5, Sept. 2006:1064-1108).

Exclusion Criteria:

* Ventricular tachyarrhythmia that may have transient or reversible causes such as: acute myocardial infarction, digitalis intoxication, drowning, electrocution, electrolyte imbalance, hypoxia, sepsis, or unstable ischemic episodes
* Incessant tachyarrhythmia
* Implanted pacemaker
* Primary disorder of bradyarrhythmia or atrial tachyarrhythmia
* Of minor age
* Pregnant
* Participating in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2006-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The percentage of patients free from complications | 6 months
Shock effectiveness for VT/VF | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Schwartz, MS, Study Director — ELA Medical, Inc.
Locations (1):
- Banner Baywood, Mesa, Arizona, United States